CLINICAL TRIAL: NCT06426212
Title: Use of Teicoplanin on a Three-weekly Administration in the Complex Outpatient Macroactivity Regimen of Infectious Diseases Unit in the Alessandro Manzoni Hospital (Lecco, Italy)
Brief Title: Use of Teicoplanin on a Three-weekly Administration in the Infectious Diseases Unit
Acronym: 3-TEICO
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Lecco (Other)
Responsible Party: Principal Investigator, Stefania Piconi, Director of Infectious Diseases Unit, Azienda Ospedaliera di Lecco
Other Study IDs: 3-TEICO
Record Dates: First submitted 2024-05-08; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Comparison of Teicoplanin Used Three Times a Week in DSIs vs NDISs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with deep infections (deep seated infections - DSIs)
  Interventions: Drug: Use of teicoplanin three times a week
- patients with superficial infections (non deep seated infections - NDSIs).
  Interventions: Drug: Use of teicoplanin three times a week

INTERVENTIONS:
Drug: Use of teicoplanin three times a week — retrospective study to evaluate the clinical effectiveness of teicoplanin therapy according to a three-weekly scheme comparing its use in the treatment of deep infections (deep seated infections - DSIs) and superficial infections (non-deep seated infections - NDSIs).

SUMMARY:
Teicoplanin is an antibiotic belonging to the class of glycopeptides, in use since 1986. Like its older "classmate" vancomycin, it inhibits protein synthesis by interfering with the synthesis of peptidoglycan, and is active on Gram-positive bacteria such as Staphilococcus spp (including MRSA), Streptococcus spp and Enterococcus spp (both faecalis and faecium).

Teicoplanin is characterized by poor gastrointestinal absorption, which requires intramuscular or intravenous administration; has a binding to plasma proteins greater than 90%; and a high volume of distribution. It reaches high levels in deep tissues (bone, abdomen, lung, kidney, heart) on the contrary it has poor penetration at the central nervous system level; it is approved for the treatment of skin and soft tissue infections, osteo-articular infections, pneumonia, endocarditis, complicated urinary tract infections, peritonitis and bacteremia associated with the aforementioned clinical conditions. Furthermore, teicoplanin has a markedly long half-life (between 30 and 180h) which allows it to be administered even every 48-72h. Dose and duration of treatment should be adjusted according to the location and severity of the infection and based on patient characteristics such as renal function. The possibility of carrying out therapeutic drug monitoring (TDM) allows maintaining plasma levels adequate for the treatment of deep infections (e.g. >20 mg/l for endocarditis) and avoiding overdose.

Thanks to the possibility of administering teicoplanin on a three-weekly schedule, patient access to hospital is further reduced.

The investigators therefore propose a retrospective study to evaluate the clinical effectiveness of teicoplanin therapy according to a three-weekly scheme by comparing its use in the treatment of deep infections (deep seated infections - DSIs) and superficial infections (non-deep seated infections - NDSIs).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Patients with documented Gram-positive infection sensitive to teicoplanin;
* Patients who have received at least 4 doses of teicoplanin on a three-weekly schedule, as monotherapy or associated with other antibiotics

Exclusion Criteria:

* Hospitalized patients
* Patients who have received less than 4 doses of teicoplanin for any cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data of patients with deep seated infections - DSIs or non deep seated infections - NDSIs treated from January 2021 to October 2023 in the Manzoni hospital in Lecco will be collected from the medical records in order to record the clinical outcomes understood as clinical resolution vs therapeutic failure, change of therapy or recurrence of infection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Describe the clinical characteristics and outcome of the study population. | 2 months
  Describe the clinical characteristics of patients and outcome (recovery vs therapeutic failure intended as death, need for modification of antibiotic therapy or recurrence of infection) of the study population.

CONTACTS AND LOCATIONS:
Locations (1):
- Stefania Piconi, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No